CLINICAL TRIAL: NCT06504771
Title: Clinical and Laboratory Patterns of Pediatric Gross Hematuria in Sohag University Hospital
Brief Title: Clinical and Laboratory Patterns of Pediatric Gross Hematuria
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Haya Mahmoud Abdelhameed, Pediatric resident at sohag general hospital, Sohag University
Other Study IDs: Soh-Med-24-06-13MS
Record Dates: First submitted 2024-07-05; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Hematuria
Keywords: Gross hematuria
MeSH Terms: conditions — Hematuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study the demographic, clinical, laboratory and etiological profile of children with gross hematuria and trace the outcome of these patients for at least 3 months follow up.

DETAILED DESCRIPTION:
Gross hematuria is a scary but common medical problem in children. This condition is considered one of the most important manifestations of kidney and urinary tract diseases. When colour of urine with blood is reddish, brown or dark or cola coloured, the condition is called as macroscopic (gross) hematuria. However, blood in urine may not always be visible to the naked eye, when it is called as microscopic hematuria.

This condition can be transient, intermittent or persistent and it may be symptomatic or asymptomatic. Hematuria originating from glomerulus is almost never bright red but usually brown, tea coloured or cola coloured. In contrary, hematuria originating from the lower urinary tract is usually pink or red in colour.

Pigments and other compounds in certain foods (including beets, berries, and food colourings) and drugs (sulfonamides, rifampicin, ibuprofen, salicylates, phenothiazines, metronidazole, phenolphthalein, chloroquine, deferoxamine, etc.) can change the colour of urine that is called false hematuria.

The causes of hematuria are very diverse, ranging from simple urinary tract infections with rapid recovery to mechanical trauma and severe glomerulonephritis with rapid decline in kidney function, it is essential to recognize the underlying disease and treat it accordingly.

The causes of gross hematuria may be categorized to whether the hematuria is glomerular or non-glomerular in origin. This distinction can be determined by microscopic examination of the urine to detect dysmorphic or monomorphic red blood cells in glomerular and non-glomerular hematuria, respectively. Although glomerular diseases are nearly always associated with some degree of hematuria, gross hematuria as a presenting manifestation is more commonly encountered with acute poststreptococcal glomerulonephritis, lupus nephritis and IgA nephropathy. Non-glomerular hematuria is most often associated with renal stones, tumours, idiopathic hypercalciuria, bacterial or viral urinary tract infection, urolithiasis and structural anomalies of the urinary tract.

It is essential to establish the cause and origin of hematuria in each case through proper history, clinical features and investigations including laboratory, radiological studies and/or percutaneous renal biopsy in some cases. But at the same time, it is important that the pediatrician is aware what any of such procedures might be helpful in establishing a proper diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* lnvestigators will include all patients complaining of gross hematuria between the ages of 1 month up to 16 years.

Exclusion Criteria:

* Children with external perineal or genital region bleeding which may falsely cause presence of blood in urine samples.
* Patients whose legal guardians will refuse participation in the study.
* Patients with follow up for less than 3 months.

Ages: 1 Month to 16 Years | Sex: All
Age Groups: Child
Study Population: patients with gross hematuria at The pediatric department and pediatric nephrology outpatient clinic at Sohag University hospital, Sohag, Egypt
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Investigate the creatinine level of the studied cases | three months
  follow up of creatinine level in mg/dl of the studied cases

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrahim Sadek, Professor, Study Director — Faculty of Medicine, Sohag university, Egypt; Ghada A Abd-Elrehim, Lecturer, Study Director — Faculty of Medicine, Sohag university, Egypt
Locations (1):
- Faculty of Medicine,Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided